CLINICAL TRIAL: NCT01552343
Title: A Double-blind, Randomized, Placebo-controlled Study Investigating the Impact Burden of Nocturia Using the Nocturia Impact Diary
Brief Title: Study Investigating the Impact Burden of Nocturia Using the Nocturia Impact Diary
Acronym: IMPACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 000034
Record Dates: First submitted 2012-03-05; First posted 2012-03-13 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Female - Desmopressin 25 μg (Experimental): Female participants took 1 tablet of 25 μg every night, approximately 1 hour prior to bedtime (with the intention to sleep), for a period of 1 month.
  Interventions: Drug: Desmopressin
- Female - Placebo (Placebo Comparator): Female participants took 1 tablet of placebo every night, approximately 1 hour prior to bedtime (with the intention to sleep), for a period of 1 month.
  Interventions: Drug: Placebo
- Male - Desmopressin 75 μg (Experimental): Male participants took 1 tablet 75 μg every night, approximately 1 hour prior to bedtime (with the intention to sleep), for a period of 1 month.
  Interventions: Drug: Desmopressin
- Male - Placebo (Placebo Comparator): Male participants took 1 tablet of placebo every night, approximately 1 hour prior to bedtime (with the intention to sleep), for a period of 1 month.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desmopressin — Desmopressin orally disintegrating tablets. Female participants took a 25 μg tablet and male participants took a 75 μg tablet one hour prior to bedtime for one month.
  Other Names: FE992026; MINIRIN®; Nocturin®
  Arms: Female - Desmopressin 25 μg; Male - Desmopressin 75 μg
Drug: Placebo — Placebo to match the 25 μg tablet of active drug taken by female participants or the 75 μg tablet taken by males. One placebo tablet taken one hour prior to bedtime for one month.
  Arms: Female - Placebo; Male - Placebo

SUMMARY:
The purpose of this study is to assess psychometric properties (reliability and validity) of the Nocturia Impact (NI) diary.

To assess the association between reduction of number of nocturnal voids and the mean changes in NI scores (sensitivity of the NI total score to change in nocturia).

To assess which NI diary items account for the main difference in change in total NI score in treatment versus placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent prior to performance of any study-related activity
2. 18 years of age (at the time of written consent) or older
3. Previous participation in FE992026 CS40 or FE992026 CS41 with a completion ≥ 30 days prior to Screening. The subject should have responded to active treatment during FE992026 CS40 or FE992026 CS41 or if he/she received placebo during these two studies he/she should have been a non-responder.
4. At least two nocturnal voids every night in two consecutive 3-day periods during the screening period (as determined by the two night-time voiding diaries dispensed at Visit 1 and collected at Visit 2)

Exclusion Criteria:

1. Chronic prostatitis (males)/chronic pelvic pain syndrome (CPPS)
2. Suspicion of bladder outlet obstruction (BOO) or a urine flow of < 5 mL/s as confirmed by uroflowmetry performed after suspicion of BOO
3. Surgical treatment, including transurethral resection, for BOO or benign prostatic hyperplasia (males) within the past six months
4. Urinary retention or a post void residual volume > 150 mL for females and > 250 mL for males as confirmed by bladder ultrasound performed after suspicion of urinary retention
5. Central or nephrogenic diabetes insipidus
6. Syndrome of inappropriate antidiuretic hormone
7. Current or a history of urologic malignancies e.g. bladder cancer
8. Genito-urinary tract pathology e.g. infection or stone in the bladder and urethra causing symptoms
9. Neurogenic detrusor activity (detrusor overactivity)
10. Suspicion or evidence of cardiac failure
11. Chronic prostatitis (males)/chronic pelvic pain syndrome (CPPS)
12. Uncontrolled hypertension
13. Uncontrolled diabetes mellitus
14. Hyponatraemia: serum sodium level must be within normal limits
15. Renal insufficiency: Serum creatinine must be within normal limits and estimated glomerular filtration rate must be ≥ 50 mL/min
16. Hepatic and/or biliary diseases: Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) levels must not be more than twice the upper limit of normal range. Total bilirubin level must not be > 1.5 mg/dL
17. History of obstructive sleep apnea
18. Treatment with another investigational product (except desmopressin) within three months prior to screening and throughout the study
19. Concomitant treatment with loop diuretics (furosemide, torsemide, ethacrynic acid)
20. Pregnancy, breastfeeding, or an intention of becoming pregnant during the period of the clinical study. Female subjects of reproductive age must have documentation of a reliable method of contraception. All pre-and perimenopausal female subjects have to perform pregnancy tests. Amenorrhea of > 12 months duration based on the reported date of the last menstrual period is sufficient documentation of post-menopausal status and does not require a pregnancy test
21. Known alcohol or substance abuse
22. Work or lifestyle that may interfere with regular night-time sleep e.g. shiftworkers 23. Any other medical condition, laboratory abnormality, psychiatric condition, mental incapacity, or language barrier which, in the judgment of the Investigator, would impair participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-03; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (10):
- United States (10):
  - South Florida Medical Research, Aventura, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Accelovance, Peoria, Illinois
  - DM Clinical Research, Springfield, Massachusetts
  - Beyer Research, Kalamazoo, Michigan
  - Remedica LLC, Rochester, Michigan
  - Accumed Research Associates, Garden City, New York
  - Radiant Research, Inc., Greer, South Carolina
  - Quality Research, Inc., San Antonio, Texas
  - Radiant Research, Inc., San Antonio, Texas

REFERENCES:
- [Result] Holm-Larsen T, Andersson F, van der Meulen E, Yankov V, Rosen RC, Norgaard JP. The Nocturia Impact Diary: a self-reported impact measure to complement the voiding diary. Value Health. 2014 Sep;17(6):696-706. doi: 10.1016/j.jval.2014.06.007. Epub 2014 Aug 20. PMID 25236993

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 67 subjects were screened and 11 subjects were screening failures: 5 due to signs of renal impairment, 4 did not have >=2 nocturnal voids every night in the 3-day screening period, 1 had uncontrolled diabetes mellitus, and 1 was leaving town for an undetermined period of time.
Groups:
- Placebo: Female and male participants took 1 tablet of placebo every night, approximately 1 hour prior to bedtime (with the intention to sleep), for a period of 1 month.
- Desmopressin: Female participants took 1 desmopressin 25 μg tablet and male participants took 1 tablet 75 μg every night, approximately 1 hour prior to bedtime (with the intention to sleep), for a period of 1 month.
Period: Overall Study
Arm/Group | Placebo | Desmopressin
Started | 29 | 27
Completed | 29 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Desmopressin | Total
Number analyzed (Participants) | 29 | 27 | 56
Age, Customized [Number; unit: participants]
  < 65 years | 11 | 13 | 24
  >=65 years | 18 | 14 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 15 | 15 | 30
Race/Ethnicity, Customized [Number; unit: participants]
  White | 25 | 23 | 48
  Black/African American | 4 | 2 | 6
  Asian | 0 | 1 | 1
  American Indian/Alaska native | 0 | 1 | 1
Ethnic Origin [Number; unit: participants]
  Hispanic or Latino | 6 | 2 | 8
  Not Hispanic or Latino | 23 | 25 | 48

OUTCOME MEASURES:

1. Primary Outcome: The Pearson Correlation Coefficient Between Change From Baseline to Month 1 in Number of Nocturnal Voids and Change From Baseline to Month 1 in Nocturia Impact (NI) Diary Total Score
Description: This outcome is a measure of sensitivity of the NI Diary to change in nocturia.
  The NI Diary is a 12-item instrument consisting of 11 core items and an overall impact question (Q12). Responses are scored from 0 (no impact) to 4 (highest impact); a lowering of score equals a decrease in impact caused by nocturia. The NI total score is the sum of the 11 core items scores. The NI total score was analyzable only if all 11 items (Q1-Q11) had non-missing responses. Otherwise, it was defined as missing. Missing values were not imputed. The average over the 3-day diary period prior to baseline (Day 1) and Month 1 was used for the overall impact score.
  The correlation was estimated using Fisher's z transformation, i.e. the NI total score was based on a standardized scale from 0 (lowest impact) to 100 (highest impact).
  Corresponding adjusted partial correlation coefficients were based on adjustments for mean number of Baseline voids, Baseline NI total score, age, and gender.
Time Frame: Day 1 (Baseline), Month 1
Population: Full analysis set. Study results are reported as per the pre-planned statistical analysis plan on combined treatment groups. The study is a psychometric evaluation of a new PRO tool and is not designed to show treatment difference between active and placebo.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Groups:
- All Participants: All study participants
Arm/Group | All Participants
Number analyzed (Participants) | 56
correlation coefficient
  Correlation - no adjustments | 0.31 [0.05 to 0.53]
  Adjusted partial correlation - baseline # of voids | 0.35 [0.09 to 0.56]
  Adj partial correlation - baseline NI total score | 0.28 [0.02 to 0.51]
  Adjusted partial correlation - age category | 0.33 [0.07 to 0.55]
  Adjusted partial correlation - gender | 0.33 [0.07 to 0.55]
Statistical Analysis 1: Comparison: All Participants; Correlation - no adjustments; Test type: Superiority or Other; p = 0.0187, t-test, 2 sided — The a priori threshold for statistical significance was 0.05
Statistical Analysis 2: Comparison: All Participants; Partial correlation - baseline # of voids; Test type: Superiority or Other; p = 0.0094, t-test, 2 sided — The a priori threshold for statistical significance was 0.05
Statistical Analysis 3: Comparison: All Participants; Partial correlation - baseline NI total score; Test type: Superiority or Other; p = 0.0383, t-test, 2 sided — The a priori threshold for statistical significance was 0.05
Statistical Analysis 4: Comparison: All Participants; Partial correlation - age category; Test type: Superiority or Other; p = 0.0133, t-test, 2 sided — The a priori threshold for statistical significance was 0.05
Statistical Analysis 5: Comparison: All Participants; Partial correlation - gender; Test type: Superiority or Other; p = 0.0128, t-test, 2 sided; The a priori threshold for statistical significance was 0.05

2. Primary Outcome: Difference in Mean Change From Baseline to Month 1 in Nocturia Impact (NI) Total Scores and Overall Impact Question for Responders and Non-Responders
Description: This outcome is a measure of sensitivity of the NI Diary to change in nocturia.
  The NI Diary is a 12-item instrument consisting of 11 core items and an overall impact question (Q12). The NI total score is defined as the sum of the 11 core items scores.
  The overall impact question (Q12) and the NI total score were transformed using Fisher's z transformation, i.e. the scores were based on a standardized scale from 0 (lowest impact) to 100 (highest impact).
  The difference in mean change in NI total score for subjects who experienced a reduction from baseline of <33% in nocturnal voids at the Month 1 visit (non-responders) versus those with a reduction in nocturnal voids from Baseline of ≥33% (responders) was estimated.
Time Frame: Day 1 (Baseline), Month 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Non-Responders: Participants who experienced a reduction from baseline of <33% in nocturnal voids at the Month 1
- Responders: Participants who experienced a reduction from baseline of >=33% in nocturnal voids at the Month 1
Arm/Group | Non-Responders | Responders
Number analyzed (Participants) | 22 | 34
units on a scale
  Nocturia Impact (NI) Total Score (Q1-Q11) | -2.6 (6.8) | -13.3 (17.9)
  Overall Impact Question (Q12) | -4.9 (15.6) | -4.9 (18.6)
Statistical Analysis 1: Comparison: Non-Responders vs Responders; Nocturia Impact (NI) Total Score (Q1-Q11); Test type: Superiority or Other; Mean Difference (Net) = 10.7, 95% CI 2-sided [2.7 to 18.8] — Non-Responders - Responders
Statistical Analysis 2: Comparison: Non-Responders vs Responders; Overall Impact Question (Q12); Test type: Superiority or Other; Mean Difference (Net) = -0.0, 95% CI 2-sided [-9.6 to 9.6] — Non-Responders - Responders

3. Primary Outcome: Cohen's D Effect Size in Responsiveness in the Nocturia Impact (NI) Total Scores and Overall Impact Question as Measured From Baseline (Day 1) to Month 1
Description: The responsiveness of the NI Diary was measured with Cohen's D effect size. The effect size was calculated for active treatment versus placebo, based on change from Baseline to Month 1. The effect size was evaluated as "small," "medium," or "large" if D was <=0.35, >0.35 - 0.65, or >0.65, respectively.
  Mean values are the Cohen's D effect size. Standard deviation is the pooled standard deviation.
Time Frame: Day 1 (Baseline), Month 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 56
units on a scale
  Nocturia Impact (NI) Total Score (Q1-Q11) | 0.73 (14.7)
  Overall Impact Question (Q12) | -0.00 (17.5)

4. Secondary Outcome: Internal Consistency of the Nocturia Impact (NI) Total Score for Each Day NI Diaries Were Completed Assessed as Cronbach's Alpha Values
Description: Cronbach's alpha (CA) is a measure of the internal consistency of the Nocturia Impact (NI) Total scores. Higher scores indicate a more reliable (precise) instrument. A value of 0.70 set as the benchmark for declaring the scale as internally consistent.
  Cronbach's alpha was assessed for each of the three consecutive days NI diaries were completed during screening (Day -20 to Day -18), baseline (Day -2 to Day 1) and Month 1 (Day 28 to Day 30).
Time Frame: Screening (Day -20 to Day -18), Baseline (Day -2 to Day 1) and Treatment (Day 28 to Day 30)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: ratio of variance
Arm/Group | All Participants
Number analyzed (Participants) | 56
ratio of variance
  Screening Day -20 | 0.915 [0.878 to 0.945]
  Screening Day -19 | 0.925 [0.892 to 0.951]
  Screening Day -18 | 0.923 [0.890 to 0.950]
  Baseline Day -2 | 0.939 [0.912 to 0.960]
  Baseline Day -1 | 0.941 [0.915 to 0.961]
  Baseline Day 1 | 0.943 [0.919 to 0.963]
  Treatment Day 28 | 0.920 [0.885 to 0.948]
  Treatment Day 29 | 0.914 [0.877 to 0.944]
  Treatment Day 30 | 0.898 [0.853 to 0.933]

5. Secondary Outcome: Construct Validity For the Nocturia Impact (NI) Total Scores and Overall Impact Question (Q12) for Participants With High/Low Number of Nocturnal Voids
Description: The known group validity was assessed by comparing participants who experienced ≥3 nocturnal voids to those who experienced <3 nocturnal voids, using the average over 3 days for the Screening and Baseline diaries. Results are reported for the NI Total Scores and the Overall Impact Question (Q12).
  The NI Diary is a 12-item instrument consisting of 11 core items and an overall impact question (Q12). The NI total score is defined as the sum of the 11 core items scores.
  The overall impact question (Q12) and the NI total score were transformed using Fisher's z transformation, i.e. the scores were based on a standardized scale from 0 (lowest impact) to 100 (highest impact).
Time Frame: Screening (Day -20), Baseline (Day 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- < 3 Voids: Study participants who had <3 voids average from the screening and baseline diaries.
- >= 3 Voids: Study participants who had >=3 voids average from the screening and baseline diaries.
Arm/Group | < 3 Voids | >= 3 Voids
Number analyzed (Participants) | 33 | 23
units on a scale
  Nocturia Impact (NI) Total Score: Screening | 28.1 (20.4) | 36.7 (23.0)
  Nocturia Impact (NI) Total Score: Baseline | 25.7 (20.4) | 39.3 (25.7)
  Overall Impact Question (Q12): Screening | 40.4 (27.3) | 56.2 (30.1)
  Overall Impact Question (Q12): Baseline | 35.6 (28.4) | 53.3 (34.7)
Statistical Analysis 1: Comparison: < 3 Voids vs >= 3 Voids; Nocturia Impact (NI) Total Score: Screening; Test type: Superiority or Other; p = 0.1471, t-test, 2 sided — The a priori threshold for statistical significance was 0.05; Mean Difference (Net) = -8.6, 95% CI 2-sided [-20.3 to 3.1]
Statistical Analysis 2: Comparison: < 3 Voids vs >= 3 Voids; Nocturia Impact (NI) Total Score: Baseline; Test type: Superiority or Other; p = 0.0318, t-test, 2 sided — The a priori threshold for statistical significance was 0.05; Mean Difference (Net) = -13.6, 95% CI 2-sided [-26.0 to -1.2]
Statistical Analysis 3: Comparison: < 3 Voids vs >= 3 Voids; Overall Impact Question (Q12): Screening; Test type: Superiority or Other; p = 0.0463, t-test, 2 sided — The a priori threshold for statistical significance was 0.05; Mean Difference (Net) = -15.8, 95% CI 2-sided [-31.2 to -0.3]
Statistical Analysis 4: Comparison: < 3 Voids vs >= 3 Voids; Overall Impact Question (Q12): Baseline; Test type: Superiority or Other; p = 0.0413, t-test, 2 sided — The a priori threshold for statistical significance was 0.05; Mean Difference (Net) = -17.7, 95% CI 2-sided [-34.6 to -0.7]

6. Secondary Outcome: Change From Baseline to Month 1 on Nocturia Impact (NI) Total Score
Description: The NI Diary is a 12-item instrument consisting of 11 core items and an overall impact question (Q12). Responses are scored from 0 (no impact) to 4 (highest impact); the NI total score is the sum of the 11 core items scores (range of 0-44) which is then transformed to a 0-100 scale (high score indicates high impact). The NI total score was analyzable only if all 11 items (Q1-Q11) had non-missing responses. Otherwise, it was defined as missing. Missing values were not imputed. The average over the 3-day diary period prior to baseline (Day 1) and Month 1 was used for the overall impact score. Negative change from baseline scores indicate a decrease in impact caused by nocturia.
Time Frame: Baseline (Day -2 to Day 1), Treatment (Day 28-30)
Population: Full analysis set. The study is a psychometric evaluation of a new PRO tool and is not designed to show treatment difference between active and placebo.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Desmopressin: Female participants took 1 tablet of 25 μg every night, approximately 1 hour prior to bedtime (with the intention to sleep), for a period of 1 month. Male participants took 1 tablet of 75 μg every night, approximately 1 hour prior to bedtime (with the intention to sleep), for a period of 1 month.
- Placebo: Participants took 1 tablet of placebo every night, approximately 1 hour prior to bedtime (with the intention to sleep), for a period of 1 month.
Arm/Group | Desmopressin | Placebo
Number analyzed (Participants) | 27 | 29
units on a scale | -8.5 (13.7) | -9.64 (17.2)
Statistical Analysis 1: Comparison: Desmopressin vs Placebo; Treatment effect. NI total scores are transformed to a 0-100 scale where 0 is good and 100 bad; Test type: Superiority; p = 0.9647, ANCOVA; Covariates baseline score, treatment and age stratum (<65, >=65); Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-6.6 to 6.3]

7. Secondary Outcome: Minimum Post-Treatment Serum Sodium Levels
Description: Serum sodium levels were monitored since hyponatremia is a potential serious adverse event associated with daily doses of desmopressin. A participant was to be withdrawn from the trial if the serum sodium level was <=125 mmol/L at any time.
Time Frame: Day 1 up to 1 month
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Female - Placebo | Male - Placebo | Female - Desmopressin 25 μg | Male - Desmopressin 75 μg
Number analyzed (Participants) | 14 | 15 | 12 | 15
participants
  <=125 mmol/L | 0 | 0 | 0 | 0
  >125 - <130 mmol/L | 0 | 0 | 0 | 0
  >=130 - 135 mmol/L | 0 | 0 | 2 | 1

8. Secondary Outcome: Summary of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: A TEAE was any adverse event occurring after start of treatment and within the time of residual drug effect, i.e. within one day of the last dose of desmopressin.
Time Frame: Day 1 up to 1 month
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Female - Placebo | Male - Placebo | Female - Desmopressin 25 μg | Male - Desmopressin 75 μg
Number analyzed (Participants) | 14 | 15 | 12 | 15
participants
  All adverse events (AEs) | 2 | 1 | 2 | 0
  Deaths | 0 | 0 | 0 | 0
  Serious AEs | 0 | 0 | 0 | 0
  AEs leading to discontinuation | 0 | 0 | 0 | 0
  Severe AEs | 0 | 0 | 0 | 0
  Adverse drug reactions (ADRs) | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Month 1
Description: A TEAE was any adverse event occurring after start of treatment and within the time of residual drug effect, i.e. within one day of the last dose of desmopressin.
Arm/Group | Placebo | Desmopressin
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/27
Other Adverse Events (participants affected / at risk) | 0/29 | 0/27

LIMITATIONS AND CAVEATS:
This was a patient reported outcome (PRO) validation study on a highly selective population (responders on active treatment and non-responsers on placebo from CS40/CS41) and not powered to look at efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.